CLINICAL TRIAL: NCT06258668
Title: Sotyktu (Deucravacitinib) Post-Marketing Surveillance in Korean Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: Real-World Safety and Effectiveness of Sotyktu (Deucravacitinib) in Patients With Moderate-to-Severe Plaque Psoriasis in Korea
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-1122
Record Dates: First submitted 2024-02-03; First posted 2024-02-14 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Moderate-to-severe Plaque Psoriasis
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed with moderate-to-severe plaque psoriasis
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — As per product label

SUMMARY:
The purpose of this observational study is to describe the safety and effectiveness of deucravacitinib in participants in Korea that have been diagnosed with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥19 years of age
* Diagnosis of moderate-to-severe plaque psoriasis
* Candidate for phototherapy or systemic therapy
* Will begin deucravacitinib according to approved product label

Exclusion Criteria:

* Participants prescribed deucravacitinib for therapeutic indications not approved in Korea
* Participants for whom deucravacitinib is contraindicated as clarified in Korean prescribing information by ministry of food and drug safety (MFDS)

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients in Korea who have been diagnosed with moderate-to-severe plaque psoriasis and have been prescribed treatment with deucravacitinib according to the approved product label.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 24 weeks from treatment initiation
Number of participants with adverse drug reactions (ADRs) | Up to 24 weeks from treatment initiation
Number of participants with serious adverse events (SAEs) | Up to 24 weeks from treatment initiation
Number of participants with serious adverse drug reactions (SADRs) | Up to 24 weeks from treatment initiation
Number of participants with unexpected adverse events (AEs) | Up to 24 weeks from treatment initiation
Number of participants with unexpected adverse drug reactions (ADRs) | Up to 24 weeks from treatment initiation
Number of participants with unexpected serious adverse events (SAEs) | Up to 24 weeks from treatment initiation
Number of participants with unexpected serious adverse drug reactions (SADRs) | Up to 24 weeks from treatment initiation

SECONDARY OUTCOMES:
Proportion of participants with static Physician Global Assessment (sPGA) of 0 or 1 | At Week 16 and/or Week 24 post treatment initiation
Number of participants achieving Psoriasis Area and Severity Index (PASI) 75 (at least a 75% improvement in PASI score from baseline) | At Week 16 and/or Week 24 post treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- South Korea (2):
  - Local Institution - 0001, Seoul
  - Novotech Laboratory Korea Co., Ltd., Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety